CLINICAL TRIAL: NCT06183411
Title: Theory of Mind in Children With DCD
Acronym: TOM_DCD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Ghent (Other)
Responsible Party: Principal Investigator, VakgroepRevalidatiewetenschappen, Prof. Dr. Lynn Bar-On, University Ghent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ONZ-2023-0329
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Developmental Coordination Disorder
Keywords: Child; Development; Theory of mind
MeSH Terms: conditions — Motor Skills Disorders | interventions — Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with DCD (Other)
  Interventions: Behavioral: Assessment

INTERVENTIONS:
Behavioral: Assessment — * Observations using two valid, observational instruments (MABC-2 and ToM test-R) that each child completes once at random.
  * A demographic and developmental questionnaire is completed once by the parent/guardian at recruitment.
  * Standardized questionnaires (Coordination Questionnaire For Parents (CVO), Social Responsiveness Scale second edition (SRS-2), Strengths and Difficulties Questionnaire (SDQ) and Theory of Mind Behavior Checklist (ToMBC)) are also questioned once to parent/guardian for data collection.

SUMMARY:
The aim of the study is to investigate theory of mind (ToM) in children with developmental coordination disorder (DCD). Dutch-speaking children, who are living in Flanders or The Netherlands (because comparisons will be made with Flemish and Dutch norms), will be included. In addition, children should be six until twelve years old with a DCD diagnosis confirmed by a multidisciplinary team (including a doctor).

During the test moment, ToM will be tested by ToM test-R and the motor skills by MABC-2. Beside, the ToM test-R will be filmed, but the child's face not shown. The parent/legal guardian will be asked to complete five online questionnaires (demographic and developmental questionnaire, CVO, SRS-2, SDQ and ToMBC), this can be completed in advance at home or at the test moment (researchers provide a laptop).

ELIGIBILITY:
Inclusion Criteria:

* Age of child: from six to 12 years old
* Confirmed diagnosis of DCD by a multidisciplinary team (including a physician)
* Child lives in Flanders or the Netherlands
* Child has Dutch as the mother tongue

Exclusion Criteria:

* Diagnosis of autism spectrum disorder (ASD)
* Blood related siblings of the child
* Parent/legal guardian does not have an adequate level of Dutch
* (IQ lower than 70) OR (no IQ information and child attends special education type 1 (mild intellectual disability) or type 2 (moderate to severe mental disability))

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Theory of Mind | 2 hours
  Measured with ToM test-R andTheory of Mind Behavior Checklist (ToMBC)

CONTACTS AND LOCATIONS:
Locations (1):
- Universiteit Gent - Vakgroep revalidatiewetenschappen, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No